CLINICAL TRIAL: NCT04139733
Title: Early Use of Prone Position in Extracorporeal Membrane Oxygenation for Severe Acute Respiratory Distress Syndrome
Brief Title: Early Use of Prone Position in ECMO for Severe ARDS
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Rui Wang, Attending doctors, Beijing Chao Yang Hospital
Other Study IDs: 2019-KE-171
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute respiratory distress syndrome; Extracorporeal Membrane Oxygenation; Prone Position
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prone group: 1. Prone position within 24 hours after VV-ECMO support.
  2. Prone position for at least 16 hours per day for a minimum of 5 days.
  Interventions: Procedure: Prone positon
- Supine group: 1. Supine group on ECMO.
  Interventions: Procedure: Supine positon

INTERVENTIONS:
Procedure: Prone positon — Prone position within 24 hours after VV-ECMO support. Prone position for at least conservative hours per day for a minimum of 5 days.
  Groups: Prone group
Procedure: Supine positon — Conventional supine position ventilation, no prone position.
  Groups: Supine group

SUMMARY:
Venovenous extracorporeal membrane oxygenation (VV-ECMO) is widely used in the salvage treatment of critical acute respiratory distress syndrome (ARDS). However, reducing lung injury, accelerating lung recovery, shortening VV-ECMO support time, and decreasing complications during the treatment need further study. By changing the body position of ARDS patients, the prone position can increase the lung's dorsal ventilation and improve the lung's ventilation/blood flow ratio to improve oxygenation. Previous multicenter studies have proved that the prone position can significantly reduce the mortality of patients with moderate and severe ARDS. However, patients with severe ARDS rescue by VV-ECMO rarely combine with a prone position.On the one hand, with the support of ECMO, the patient's oxygenation will be significantly improved, and they will no longer need the assistance of a prone position. In addition, the ECMO cannula brings some challenges to implementing a prone position. Only a few cohort studies have reported that VV-ECMO combined with a prone position could improve the oxygenation index and respiratory system compliance during the late treatment period.

The initial reason for PP in ARDS patients was to alleviate severe hypoxemia, as it was an efficient means to improve oxygenation in most patients. However, some patients were categorized as non-responders in the PP regarding oxygenation, which caused VV-ECMO therapy to be initiated. Should we decide to perform PP after VV-ECMO therapy no longer? This study evaluates whether early use of PP during VV-ECMO would increase the proportion of patients successfully weaned from VV-ECMO support compared with supine positioning in severe ARDS patients who received PP before ECMO.

ELIGIBILITY:
Inclusion Criteria:

1. met the diagnostic criteria of Berlin's definition for ARDS;
2. had undergone prone positing before VV-ECMO；
3. receiving VV-ECMO support

Exclusion Criteria:

1. spinal instability；
2. elevated intracranial pressure;
3. facial/neck trauma;
4. recent sternotomy;
5. large ventral surface burn;
6. multiple trauma with unstabilized fractures;
7. severe hemodynamic instability;
8. massive hemoptysis;
9. high risk of requiring CPR or defibrillation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had undergone PP as rescue therapy before VV-ECMO
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
The proportion of patients successfully weaned from VV-ECMO, | After patients enrolled 60 days
  Weaning VV-ECMO more than 48 hours with stable oxygenation and no need to re-establish ECMO

SECONDARY OUTCOMES:
60-day mortality | After patients enrolled 60 days
  Mortality rate at 60 days of VV-ECMO support

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, Dr., Principal Investigator — Beijing Chao-Yang Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Combes A, Hajage D, Capellier G, Demoule A, Lavoue S, Guervilly C, Da Silva D, Zafrani L, Tirot P, Veber B, Maury E, Levy B, Cohen Y, Richard C, Kalfon P, Bouadma L, Mehdaoui H, Beduneau G, Lebreton G, Brochard L, Ferguson ND, Fan E, Slutsky AS, Brodie D, Mercat A; EOLIA Trial Group, REVA, and ECMONet. Extracorporeal Membrane Oxygenation for Severe Acute Respiratory Distress Syndrome. N Engl J Med. 2018 May 24;378(21):1965-1975. doi: 10.1056/NEJMoa1800385. PMID 29791822
- [Background] Scholten EL, Beitler JR, Prisk GK, Malhotra A. Treatment of ARDS With Prone Positioning. Chest. 2017 Jan;151(1):215-224. doi: 10.1016/j.chest.2016.06.032. Epub 2016 Jul 8. PMID 27400909
- [Background] Fernandez R, Trenchs X, Klamburg J, Castedo J, Serrano JM, Besso G, Tirapu JP, Santos A, Mas A, Parraga M, Jubert P, Frutos F, Anon JM, Garcia M, Rodriguez F, Yebenes JC, Lopez MJ. Prone positioning in acute respiratory distress syndrome: a multicenter randomized clinical trial. Intensive Care Med. 2008 Aug;34(8):1487-91. doi: 10.1007/s00134-008-1119-3. Epub 2008 Apr 22. PMID 18427774
- [Background] Taccone P, Pesenti A, Latini R, Polli F, Vagginelli F, Mietto C, Caspani L, Raimondi F, Bordone G, Iapichino G, Mancebo J, Guerin C, Ayzac L, Blanch L, Fumagalli R, Tognoni G, Gattinoni L; Prone-Supine II Study Group. Prone positioning in patients with moderate and severe acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2009 Nov 11;302(18):1977-84. doi: 10.1001/jama.2009.1614. PMID 19903918
- [Background] Sud S, Friedrich JO, Taccone P, Polli F, Adhikari NK, Latini R, Pesenti A, Guerin C, Mancebo J, Curley MA, Fernandez R, Chan MC, Beuret P, Voggenreiter G, Sud M, Tognoni G, Gattinoni L. Prone ventilation reduces mortality in patients with acute respiratory failure and severe hypoxemia: systematic review and meta-analysis. Intensive Care Med. 2010 Apr;36(4):585-99. doi: 10.1007/s00134-009-1748-1. Epub 2010 Feb 4. PMID 20130832
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Reutershan J, Schmitt A, Dietz K, Unertl K, Fretschner R. Alveolar recruitment during prone position: time matters. Clin Sci (Lond). 2006 Jun;110(6):655-63. doi: 10.1042/CS20050337. PMID 16451123
- [Background] Lee JM, Bae W, Lee YJ, Cho YJ. The efficacy and safety of prone positional ventilation in acute respiratory distress syndrome: updated study-level meta-analysis of 11 randomized controlled trials. Crit Care Med. 2014 May;42(5):1252-62. doi: 10.1097/CCM.0000000000000122. PMID 24368348
- [Background] Kimmoun A, Roche S, Bridey C, Vanhuyse F, Fay R, Girerd N, Mandry D, Levy B. Prolonged prone positioning under VV-ECMO is safe and improves oxygenation and respiratory compliance. Ann Intensive Care. 2015 Dec;5(1):35. doi: 10.1186/s13613-015-0078-4. Epub 2015 Nov 4. PMID 26538308
- [Background] Guervilly C, Hraiech S, Gariboldi V, Xeridat F, Dizier S, Toesca R, Forel JM, Adda M, Grisoli D, Collart F, Roch A, Papazian L. Prone positioning during veno-venous extracorporeal membrane oxygenation for severe acute respiratory distress syndrome in adults. Minerva Anestesiol. 2014 Mar;80(3):307-13. Epub 2013 Nov 21. PMID 24257150
- [Background] Kipping V, Weber-Carstens S, Lojewski C, Feldmann P, Rydlewski A, Boemke W, Spies C, Kastrup M, Kaisers UX, Wernecke KD, Deja M. Prone position during ECMO is safe and improves oxygenation. Int J Artif Organs. 2013 Nov;36(11):821-32. doi: 10.5301/ijao.5000254. Epub 2013 Oct 2. PMID 24338657
- [Background] Culbreth RE, Goodfellow LT. Complications of Prone Positioning During Extracorporeal Membrane Oxygenation for Respiratory Failure: A Systematic Review. Respir Care. 2016 Feb;61(2):249-54. doi: 10.4187/respcare.03882. Epub 2015 Oct 13. PMID 26464520
- [Derived] Wang R, Tang X, Li X, Li Y, Liu Y, Li T, Zhao Y, Wang L, Li H, Li M, Li H, Tong Z, Sun B. Early reapplication of prone position during venovenous ECMO for acute respiratory distress syndrome: a prospective observational study and propensity-matched analysis. Ann Intensive Care. 2024 Aug 20;14(1):127. doi: 10.1186/s13613-024-01365-4. PMID 39162882
- [Derived] Petit M, Fetita C, Gaudemer A, Treluyer L, Lebreton G, Franchineau G, Hekimian G, Chommeloux J, Pineton de Chambrun M, Brechot N, Luyt CE, Combes A, Schmidt M. Prone-Positioning for Severe Acute Respiratory Distress Syndrome Requiring Extracorporeal Membrane Oxygenation. Crit Care Med. 2022 Feb 1;50(2):264-274. doi: 10.1097/CCM.0000000000005145. PMID 34259655